CLINICAL TRIAL: NCT01799317
Title: Regulation of Bone Mineralization in Renal Osteodystrophy
Brief Title: How Bone is Made in Children Receiving Dialysis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of California, Los Angeles (Other)
Collaborators: Children's Hospital Los Angeles (Other); Loma Linda University (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Isidro Salusky, MD, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: IBS-05; R01DK035423-19 (NIH)
Record Dates: First submitted 2013-02-20; First posted 2013-02-26 (Estimated); Last update posted 2013-02-26 (Estimated); Status verified 2013-02

CONDITIONS: Bone Mineralization Defect
MeSH Terms: interventions — Ergocalciferols

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment with vitamin D2 (Active Comparator): Vitamin D2 50,000u titrated to serum 25(OH)D values given orally once a month in addition to standard of care: Doxercalciferol escalating doses beginning at 2.5 mcg given orally thrice weekly. Sevelamer Carbonate 800 mg (1600- 4800 mg) given orally with each meal
  Interventions: Drug: Vitamin D2
- Standard of Care (No Intervention): Standard of Care: Doxercalciferol escalating doses beginning at 2.5 mcg given orally thrice weekly. Sevelamer Carbonate 800 mg (1600- 4800 mg) given orally with each meal

INTERVENTIONS:
Drug: Vitamin D2 — These patients will receive standard of care vitamin D 1,25 therapy with intervention of vitamin D2
  Other Names: Ergocalciferol
  Arms: Treatment with vitamin D2

SUMMARY:
The study outlined is designed to measure and to determine whether the combined use of vitamin D2 (ergocalciferoI) and 1-alpha-hydroxyvitamin D2 (doxercalciferol)) or doxercalciferol alone will correct the mineralization defect in pediatric patients with established secondary hyperparathyroidism (2°HPT) undergoing regular peritoneal dialysis. Serum phosphorus levels will be controlled with a calcium¬-free-metal free phosphate binder; (obtained at baseline and after 8 months of treatment) sevelamer. Indices of bone mineralization obtained at baseline and after 8 months of treatment will be measured by quantitative histomorphometry in iliac crest bone biopsies after double tetracycline labeling. Immunohistochemistry will be done in specimens of bone biopsies from iliac crest to examine the expression for selected markers of bone turnover and mineralization such as FGF-23, DMP1, MEPE and OPG. Serum PTH levels will be measured with the 1st and 2nd generation immunometric assay (PTH-IMAs) and fibroblast growth factor-23 (FGF-23) will be determined by one assay with specific detection antibodies that are against epitopes within the C-terminus of FGF-23 and another assay that uses antibodies against epitopes within the N- and C-terminal portions of the molecule respectively. The value of non-invasive assessment of bone mass by quantitative computed tomography (QCT) and its relationship with vascular disease determined by ultrasound (US) of intimal carotid thickness (CIMT) will be correlated with bone histomorphometry and the different biochemical determinations.

ELIGIBILITY:
Inclusion Criteria:

* medically stable patients
* 6-21 years old
* undergoing treatment with continuous cycling peritoneal dialysis
* evidence of mineralization defect and secondary hyperparathyroidism

Exclusion Criteria:

* histopathological lesion of bone such as adynamic bone or osteomalacia
* poor compliance
* current treatment with prednisone or other immunosuppressives
* treatment with human recombinant growth hormone
* parathyroidectomy

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-03; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Improvement of bone mineralization defect demonstrated by bone histomorphometry | 8 months
  Iliac crest bone biopsy pre and post treatment with vitamin D2

SECONDARY OUTCOMES:
Radiographic improvement of skeletal abnormalities associated with renal osteodystrophy | 8 months
  We will compare skeletal lesions identified through radiographic studies with bone histomorphometry pre and post treatment with vitamin D2

CONTACTS AND LOCATIONS:
Overall Officials: Isidro Salusky, MD, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - Loma Linda University, Loma Linda, California
  - Childrens Hospital Los Angeles, Los Angeles, California